CLINICAL TRIAL: NCT00035581
Title: A Multi-Center, Randomized, Controlled Study of the Biological Actions of Ampligen as an Adjunct to HAART in HIV Disease
Brief Title: Safety and Efficacy of Ampligen in the Treatment of HIV Patients Failing HAART
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: AIM ImmunoTech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMP 719
Record Dates: First submitted 2002-05-03; First posted 2002-05-06 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: HIV Seropositivity; HIV Infection
Keywords: treatment experienced; HIV Infections; HIV; HAART; early virologic failure
MeSH Terms: conditions — HIV Seropositivity; HIV Infections | interventions — poly(I).poly(c12,U)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ampligen (Experimental): Ampligen (polyI-polyC12U) 200-400 mg IV infusions given twice weekly for 24 weeks
  Interventions: Drug: poly I-poly C12U
- No Ampligen (No Intervention): No Ampligen administered for first 24 weeks

INTERVENTIONS:
Drug: poly I-poly C12U — 200-400 mg IV infusions 2x/week for 24 weeks
  Other Names: Ampligen; Rintatolimod
  Arms: Ampligen

SUMMARY:
This is an open-label, prospective, randomized, controlled study of the safety and efficacy including clinical, immunologic, and virologic assessments of adding Ampligen to "HAART" in HIV infected patients with CD4 counts >300 and HIV-1 plasma RNA >500 and <30,000 copies/ml (PCR).

ELIGIBILITY:
1. Adults at least 18 years of age.
2. CD4 cell count of >300 cells.
3. HIV-1 plasma RNA >500 and <30,000 copies/ml.

   A qualifying ("screening") HIV-1 RNA level >500 and <30,000 copies/ml must be documented at least once within 40 days prior to starting Baseline while patient is receiving a HAART regimen containing at least two of the following antiretroviral drugs:
   * Abacavir (Ziagen)
   * Zidovudine (Retrovir) AZT
   * Zalcitabine (Hivid) ddC
   * Didanosine (Videx) ddI
   * Stavudine (Zerit) d4T
   * Efavirenz (Sustiva)
   * Indinavir (Crixivan)
   * Ritonavir (Norvir)
   * Nelfinavir (Viracept)
   * Amprenavir (Agenerase)

   The patient must have been taking this HAART regimen for four months or longer at the time of the qualifying HIV-1 RNA determination.
4. History of prior treatment (including the current HAART regimen) with at least one protease inhibitor (PI) and at least two nucleoside reverse transcriptase inhibitors (NRTI) and/or at least one non-nucleoside reverse transcriptase inhibitor (NNRTI) and at least two nucleoside reverse transcriptase inhibitors (NRTI).
5. Karnofsky performance status of at least 70.
6. The following laboratory parameters within 14 days prior to treatment:

   * Hemoglobin > 9.2 g/dL for men and > 8.9 g/dL for women
   * Neutrophil count > 1000
   * Platelet count > 75,000
   * AST/ALT < 4.0 x upper limit of normal (ULN)
   * Serum creatinine < 1.5 x ULN or a creatinine clearance > 50 mL/min.
7. For females with child bearing potential: A negative serum pregnancy test within 14 days prior to randomization. Males and females of child bearing potential agree to use an effective means of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2001-05; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Reduction in HIV-1 Viral Load | 4, 8, 12, 16, 20 and 24
  Evaluate the effects of adding Ampligen (or no Ampligen) to "HAART" in HIV+ patients for evidence of reductions in HIV-1 viral load in plasma using Roche Amplicor assay.

CONTACTS AND LOCATIONS:
Overall Officials: David R Strayer, MD, Study Director — AIM ImmunoTech Inc.
Locations (7):
- United States (7):
  - Orange County Center for Special Immunology, Fountain Valley, California
  - Circle Medical Center, Norwalk, Connecticut
  - Dupont Circle Physicians Group, Washington D.C., District of Columbia
  - Julia Torres, MD, Fort Lauderdale, Florida
  - Scott Ubillos, MD, Tampa, Florida
  - St. Michael's Medical Center, Newark, New Jersey
  - W. Chris Woodward, DO, Reading, Pennsylvania